CLINICAL TRIAL: NCT04639024
Title: An Open-label Pilot Study to Evaluate the Safety and Efficacy of ADCT-301 in Patients With Relapsed or Refractory Acute Myeloid Leukemia, Myelodysplastic Syndrome, or Myeloproliferative Neoplasms.
Brief Title: ADCT-301 in Patients With R/R AML, MDS, or MDS/MPN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: ADCT is reallocating all resources to the phase III program.
Sponsor: Gwynn Long, M.D. (Other)
Collaborators: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor-Investigator, Gwynn Long, M.D., Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105771
Record Dates: First submitted 2020-11-05; First posted 2020-11-20 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Myeloproliferative Neoplasm (MDS/MPN)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADCT-301 Infusion (Experimental): Patients will receive ADCT-301 37.5 ug/kg infused day 1,8, and 15 of a q3week cycle. Patients will have up to 2 cycles to assess response and safety to therapy and if they are not progressing may continue for up to 6 cycles.
  Interventions: Drug: ADCT-301

INTERVENTIONS:
Drug: ADCT-301 — Patients will receive ADCT-301 37.5 ug/kg infused day 1,8, and 15 of a q3week cycle. Patients will have up to 2 cycles to assess response and safety to therapy and if they are not progressing may continue for up to 6 cycles.
  Other Names: Camidanlumab tesirine

SUMMARY:
This is research study to find out if a drug called ADCT-301 is safe and to look at how patients respond to the study drug after an allogeneic transplantation.

ADCT-301 will be administered on Days 1, 8 and 15 with blood tests following study drug infusion. Patients will have a bone marrow biopsy at the end of cycle 2/before cycle 3 to see how they are responding to the study drug.

Patients will be followed for approximately every 12 weeks from the last disease assessment for up to 1 year from completion of therapy.

There are risks to this study drug. Some risks include: decrease in certain blood cells, weight loss, loss of appetite, rash and Guillain-Barre syndrome, where the immune system attacks and damages nerves.

ELIGIBILITY:
Inclusion Criteria:

Patients ≧ 18 years of age with persistence or relapse/progression AML, MDS, or MDS/MPN,

1. following allogeneic stem cell transplantation.

   * grade 1 overall GVHD at time of inclusion with stable immune suppression for at least 2 weeks pre infusion on study and planned stable immune suppression dose for at least 8 weeks (the safety evaluation period)
2. Calculated creatinine clearance ≥ 60ml/min as estimated by Cockcroft Gault and not dialysis dependent.
3. AST, ALT <3 x ULN unless documented due to medications (ie azole or other common therapy for such patients). Total bilirubin ≤3.0 mg/dl unless there is a history of Gilbert's syndrome in which case the T bili hould be < 5.0 mg/dl.
4. Females cannot be pregnant or breast-feeding from time of enrollment till 16 weeks post final agent exposure on this study.
5. Immune suppression not greater than 20mg prednisone daily or equivalent dosing of alternative GVHD prophylaxis/therapy
6. Patients are at least 30 days from most recent allogeneic stem cell infusion
7. Patients may have had other therapy post alloBMT and other donor lymphocyte infusions but they must be at least 60 days from the last infusion of cell therapy products
8. Patients must have other anti-leukemia therapies stopped 2 weeks prior to infusion on this study. Hydrea or pheresis ARE allowed prior to this study and may continue until 14 days following the first infusion on this study if deemed to be needed to assist in count control.

Exclusion Criteria:

1. Patients with progressive infections at time of first infusion (patients with treated infections documented as controlled by the treating team are eligible).
2. Known active CNS disease at time of enrollment
3. Patients with other cancers treated within 3 years
4. Known history of immunogenicity or hypersensitivity to a CD25 antibody or a component of ADCT-301
5. Major surgery, chemotherapy, systemic therapy (excluding hydroxyurea, steroids, and any targeted small molecules or biologics), or radiotherapy within 14 days or 5 half-lives (whichever is shorter) prior to Cycle 1, Day 1 treatment, except if approved by Dr. Rizzieri.
6. Patients with proven, progressive severe autoimmune disease such as multiple sclerosis, active Guillain Barré syndrome, poliomyelitis, sjogren's are not eligible. Given the immediate, life threatening nature of the relapsed cancer in this patient population, those with other stable and non-immediate non-threatening autoimmune disorders such as thyroid disease or diabetes and others are eligible.
7. Patients with a known infection/reactivation of any of the following within 28 days of the first dose of this agent on study are not eligible: HSV1, HSV2, VZV, EBV, CMV, measles, influenza A, Zika, Chikungunya, mycoplasma pneumonia, Campylobacter jejuni, enterovirus B68, or SARS-CoV-2. Patients will have evaluation for HSV1, HSV2, VZV, EBV, CMV as part of screening studies. Patients will have SARS-CoV-2 screening performed if at all possible during the screening process. If screening is not available, then screening based on symptoms will be documented. Additionally, screening based on clinical concern and/or symptoms will be conducted for measles, influenza A, Zika, Chikungunya, mycoplasma pneumonia, Campylobacter jejuni, enterovirus B68.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Morphologic complete response rate of ADCT-301 | End of Study, up to 3 years
  Investigator report; efficacy rule
Safety of ADCT-301 | up to 12 weeks (84 days) after the last dose
  Number of adverse events as measured by self report

CONTACTS AND LOCATIONS:
Overall Officials: Gwynn Long, M.D., Principal Investigator — Professor of Medicine
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No